CLINICAL TRIAL: NCT02005692
Title: A Pilot Study to Assess the DynaSense System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leaf Healthcare, Inc. (Industry)
Collaborators: Centauri Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CM-002
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Pressure Ulcers
Keywords: pressure ulcers; bed sores; patient turn protocol; patient movement; patient monitoring
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- DynaSense sensor (Experimental)
  Interventions: Device: DynaSense sensor

INTERVENTIONS:
Device: DynaSense sensor

SUMMARY:
The study is designed to test the DynaSense system, which is a patient movement and orientation monitoring system. The study is intended to determine that:

* the DynaSense system identifies patients that are not turning adequately on their own and therefore require caregiver-assisted turns.
* the DynaSense system identifies patients that are turning adequately on their own and therefore do not require a caregiver-assisted turn.
* the DynaSense system helps ensure compliance with an institution's established patient turning protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female 18 to 110 years of age;
* Inpatient currently on the unit and expected to remain for at least 12 hours;
* Able and willing to comply with the study procedures;
* Subject (or his/her agent) is able to read, understand, and provide Informed Consent in the English language.

Exclusion Criteria:

* Subject is a female subject under the age of 60 who is pregnant, planning on becoming pregnant, or is currently breastfeeding.

  1. Any woman under the age of 60, must have a negative urine pregnancy test prior to being enrolled in the study; OR
  2. Be postmenopausal for at least 2 years, OR
  3. have had a bilateral tubal ligations, OR
  4. have had a bilateral oophorectomy, OR
  5. have had a hysterectomy.
* Subjects with a known tape allergy or sensitivity to EKG leads or similar types of adhesives used in common medical products.
* Subjects who cannot have the patient sensor applied on the surface of the patient's anterior torso.
* Subjects who have a pacemaker or implantable cardiovascular-defibrillator (ICD).
* Subjects with dementia, Alzheimer's disease or other mental disabilities and incapacitation that would prevent the subject from providing written informed consent. If the subject is unable to provide informed consent due to mental incapacity, then the subject's Durable Power of Attorney may provide informed consent and sign the informed consent on behalf of the subject.
* Subjects who refuse to have an area of hair on their chest be clipped or shaved, if needed for patient sensor adhesion.
* Subjects, who in the opinion of the Principal Investigator, are at increased risk by participating in the clinical study.
* Subjects who have participated in another clinical study within the past 30 days or are currently participating in another clinical study at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Pezzani, MD, Principal Investigator — El Camino Hospital
Locations (1):
- El Camino Hospital, Mountain View, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DynaSense Sensor: All patients enrolled in the study were prescribed a Q2 hour (every 2 hour) turning protocol, as per the standard guidelines of the study site. In the context of the study, caregivers were not asked to turn patients any more or less frequently than what the study site's standard turning protocol required.
  The rate of compliance with prescribed turning protocols was measured using the DynaSense System.
Period: Overall Study
Arm/Group | DynaSense Sensor
Started | 70
Completed | 63
Not Completed | 7
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Discharged earlier than anticipated | 5

BASELINE CHARACTERISTICS:
Population: All subjects who successfully completed the study.
Groups:
- DynaSense Sensor: All subjects who successfully completed the study.
Arm/Group | DynaSense Sensor
Number analyzed (Participants) | 63
Age, Continuous [Mean (Full Range); unit: years] | 63 [23 to 97]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Safety Primary Endpoint
Description: The safety primary endpoint is to assess safety by documenting the number, type, and severity of side effects and adverse events.
Time Frame: Subjects will be followed for the length of hospital stay which is expected to average 5 days, or until resolution of ADE.
Measure: Number; unit: percentage of subjects with ADEs
Groups:
- DynaSense Sensor: All subjects enrolled in the study.
Arm/Group | DynaSense Sensor
Number analyzed (Participants) | 70
percentage of subjects with ADEs | 2.86

2. Primary Outcome: Turn Protocol Compliance
Description: The primary clinical efficacy endpoint is to assess the change in turning protocol compliance after implementation of the DynaSense system.
Time Frame: Subjects will be followed for the length of hospital stay which is expected to average 5 days.
Measure: Number (95% Confidence Interval); unit: percentage turn compliance
Arm/Group | DynaSense Sensor
Number analyzed (Participants) | 63
percentage turn compliance | 98 [97 to 99]

ADVERSE EVENTS:
Time Frame: Upon removal of the patient sensor (within 5 minutes of removal), the subject's skin was assessed for any ADEs.
Description: If an ADE was present upon sensor removal, the subject's skin was re-assessed approximately 1 hour later prior to hospital discharge when possible. If re-assessment was not possible prior to discharge, a follow-up telephone call was made to subjects to determine time to resolution.
Arm/Group | DynaSense Sensor
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 2/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DynaSense Sensor (N=70)
Erythema (Skin Redness) (Skin and subcutaneous tissue disorders) | 1 (1) — Localized erythema (skin redness) following removal of patient sensor.
Itching (Skin and subcutaneous tissue disorders) | 1 (1) — Localized itching in skin region where patient sensor was removed.
Skin Irritation/Discomfort (Skin and subcutaneous tissue disorders) | 2 (2) — Skin irritation and discomfort following removal of patient sensor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less